CLINICAL TRIAL: NCT02803892
Title: Evaluation of the Efficacy of Rapamycin and a Dipeptidyl Peptidase-4 Inhibitor (Vildagliptin) in Improving Beta Cell Function in Type 1 Diabetes of Long Duration, a Perspective Randomized Study
Brief Title: Monotherapy With Rapamycin in Long-standing Type 1 Diabetes
Acronym: MONORAPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Piemonti Lorenzo (Other)
Collaborators: Italian Diabetes Foundation (Other)
Responsible Party: Sponsor-Investigator, Piemonti Lorenzo, Director San Raffaele Diabetes Research Institute (SR-DRI), Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI-2/2014 MONORAPA
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sirolimus; Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Group 1: Placebo (Placebo Comparator): Eligible participants will be randomized to one of three treatment arms. In this arm patients will received placebo x 2 placebo (Group 1) After 4 weeks of treatment, patients will discontinue relevant placebo treatment, but continue the second placebo for a further 8 weeks
  Interventions: Drug: Placebo 1; Drug: Placebo 2
- Group 2: Rapamycin plus Placebo (Experimental): Eligible participants will be randomized to one of three treatment arms. In this arm patients will received rapamycin plus placebo. After 4 weeks of treatment, patients will discontinue rapamycin, but continue the second placebo for a further 8 weeks
  Interventions: Drug: rapamycin; Drug: Vildagliptin
- Group 3: Rapamycin plus Vildagliptin (Experimental): Eligible participants will be randomized to one of three treatment arms. In this arm patients will received rapamycin plus vildagliptin. After 4 weeks of treatment, patients will discontinue rapamycin , but continue Vildagliptin o for a further 8 weeks
  Interventions: Drug: rapamycin; Drug: Vildagliptin

INTERVENTIONS:
Drug: rapamycin — Rapamycin will be administered at an initial dose 0.2 mg/kg on day 0, followed by 0.1 mg/kg/die. The daily dose will be adjusted to the whole blood 24-hr trough to target, as tolerated, 8-10 ng/mL
  Other Names: Rapamune®
  Arms: Group 2: Rapamycin plus Placebo; Group 3: Rapamycin plus Vildagliptin
Drug: Vildagliptin — Vildagliptin will be administered at a dose of 50 mg x2/die starting from day 0.
  Other Names: GALVUS
  Arms: Group 2: Rapamycin plus Placebo; Group 3: Rapamycin plus Vildagliptin
Drug: Placebo 1 — Placebo 1 will be titrated according to a random schedule alternating plausible doses of placebo. After 4 weeks of treatment patients will discontinue placebo 1
  Arms: Group 1: Placebo
Drug: Placebo 2 — Placebo 2 will be administered BID starting from day 0. After 8 weeks of treatment patients will discontinue placebo 2
  Arms: Group 1: Placebo

SUMMARY:
This study is a phase 2, single-center, prospective, randomized, double-blind, placebo-controlled, 3-arm parallel group (1:1:1) intervention trial to determine the efficacy of 4 weeks rapamycin treatment and 4 weeks rapamycin treatment plus 3 months vildagliptin treatment versus placebo in increasing endogenous insulin production and correcting glycemic lability. It will involve 60 patients with long standing type 1 diabetes (T1D). Patients will receive for one month placebo (Group 1), rapamycin plus placebo (Group 2), or rapamycin plus Vildagliptin (Group 3). Rapamycin will be administered at an initial dose 0.2 mg/kg orally on day 0 followed by 0.1 mg/kg/die (target trough levels: 8-10 ng/ml). Vildagliptin will be administered at a dose of 50 mg x2/die starting from day 0. After 4 weeks of treatment (period A), patients will discontinue rapamycin or relevant placebo treatment, but continue Vildagliptin or placebo for a further 8 weeks and be monitored over this period (period B).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >18 years, inclusive
* Clinical history compatible with T1D with onset of disease at < 40 years of age, insulin dependence for ≥ 5 years at the time of enrolment
* C-peptide concentrations under the threshold of preserved beta cell function: fasting C peptide <0.23 ng/ml
* Detectable fasting proinsulin concentrations (>0.5 pmol/l)
* Ability to provide written informed consent
* Mentally stable and able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations

Exclusion Criteria:

* Body mass index (BMI) >30 kg/m2 or patient with body weight ≤40kg;
* Insulin requirement >1.0 IU/kg/day or <10 U/day;
* HbA1c >11% (normal value: 3.5-6.0%) at the time of enrolment
* estimated glomerular filtration rate <60 mL/min/1.73m2 calculated using the subject's measured serum creatinine and the Modification of Diet in Renal Disease [MDRD] study estimation formula)
* Presence or history of macroalbuminuria (>300mg/g creatinine)
* For female subjects: positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation of treatment
* Active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB) as determined by a positive skin test or clinical presentation, or under treatment for suspected TB
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Lymphopenia (<1,000/μL), neutropenia (<1,500/μL), or thrombocytopenia (platelets <100,000/μL).
* Severe unremitting diarrhea, vomiting or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications
* Any medical condition that will interfere with safe participation in the trial;
* Any immunosuppressive treatment at the time of enrollment.
* Allergy to active ingredients or to any of excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline C-peptide response in the MMTT | week 4±1, week 12±2
  the proportion of participants with a positive response to the MMTT defined as C-peptide at 90 min >0.6 ng/ml.
Change from Baseline C-peptide after the MMTT | week 4±1, week 12±2
  change in the area under the curve of C-peptide after the MMTT vs baseline

SECONDARY OUTCOMES:
Change from Baseline insulin requirement | week 4±1, week 12±2
  change in insulin requirement vs baseline
Change from Baseline fasting C-peptide | week 4±1, week 12±2
  change in fasting C-peptide vs baseline
Change from Baseline HbA1c | week 4±1, week 12±2
  change in HbA1c vs baseline
Adverse Events (AEs) related to the immunosuppression | week 4±1, week 12±2
  the incidence and severity of Adverse Events (AEs) related to the immunosuppressive treatment
Adverse Events (AEs) and Serious Adverse Events (SAEs) | week 4±1, week 12±2
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Ospedale San Raffaele; Emanuele Bosi, MD, Study Chair — Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Bolla AM, Gandolfi A, Borgonovo E, Laurenzi A, Caretto A, Molinari C, Catalano RS, Bianconi E, Monti P, Sordi V, Pellegrini S, Lampasona V, Costa S, Scavini M, Bosi E, Piemonti L. Rapamycin Plus Vildagliptin to Recover beta-Cell Function in Long-Standing Type 1 Diabetes: A Double-Blind, Randomized Trial. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e507-e519. doi: 10.1210/clinem/dgaa791. PMID 33124663